CLINICAL TRIAL: NCT00452140
Title: Phase II Study for Repeated Dosing of the Trifunctional Bispecific Anti-HER-2/Neu x Anti-CD3 Antibody Ertumaxomab in Patients With HER-2/Neu 1+ or 2+/FISH Negative Expressing Advanced or Metastatic Breast Cancer (Stage IIIb/IV) Progressing After Endocrine Treatment
Brief Title: Phase II Study With the Trifunctional Antibody Ertumaxomab to Treat Metastatic Breast Cancer Progressing After Endocrine Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: company focus on other projects
Sponsor: Neovii Biotech (Industry)
Responsible Party: Fresenius Biotech GmbH, Fresenius Biotech GmbH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IV-ERT-BC-03; EudraT number: 2006-005017-36
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Metastatic Breast Cancer; Advanced Breast Cancer
Keywords: Breast Cancer; investigational drug; drug therapy; Antineoplastic Protocols; Immunotherapy; Metastatic breast cancer; Advanced breast cancer; Stage III to IV breast cancer; Hormonal therapy refractory; Failure of hormonal therapy; Her-2/neu expressing breast cancer; Her-2/neu
MeSH Terms: conditions — Breast Neoplasms | interventions — ertumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: ertumaxomab — 10 µg, IV on day 0 followed by 100 µg every 7 days up to a maximum of 12 infusions.

SUMMARY:
The purpose of the study is to demonstrate clinical efficacy of the investigational trifunctional bispecific antibody ertumaxomab for treatment of patients with HER-2/neu 1+ or 2+ (FISH-) expressing advanced or metastatic breast cancer (stage III b/IV) which has progressed after endocrine therapy.

Ertumaxomab is a trifunctional bispecific antibody targeting Her-2/neu and CD3 on T cells. Trifunctional antibodies represent a new concept for targeted anticancer therapy. This new antibody class has the capability to redirect T cells and accessory cells (e.g. macrophages, dendritic cells [DCs] and natural killer [NK] cells) to the tumor site. According to preclinical data, trifunctional antibodies activate these immune cells, which can trigger a complex anti-tumor immune response.

DETAILED DESCRIPTION:
An open-label, non-randomized, uncontrolled, one-stage, phase II study evaluating the efficacy and safety of the investigational trifunctional bispecific antibody ertumaxomab (anti-Her-2/neu x anti-CD3) for the treatment of hormone therapy refractory advanced or metastatic breast cancer tumours (stage IIIb or IV) which are known to express HER-2/neu (1+ or 2+/FISH negative).Ertumaxomab will be administered at 7 day intervals by constant rate 3 hour intravenous (i.v.) infusions according to the following sequential dose schedule: 10 µg (day 0) and thereafter 100 µg flat doses once every 7 days (± 1 day) for a maximum of up to 12 weeks or until disease progression or any other unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Women ≥ 18 years, negative pregnancy test at screening life expectancy of at least 6 months
* Locally advanced (stage IIIb) or metastatic (stage IV) and not curable adenocarcinoma of the breast
* Measurable disease, defined as at least one lesion that is measurable in one dimension (RECIST)
* HER-2/neu expression 1+ or 2+ / FISH negative
* Estrogen Receptors (ERs) and/or Progesterone Receptors (PRs) positive
* Prior adequate endocrine therapy for advanced or metastatic disease
* Disease progression during or after endocrine therapy
* No prior treatment with mouse or rat antibodies
* ECOG performance score of ≤ 1
* Adequate hematological, liver and kidney function

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Known HIV infection or Presence of autoimmune disease or other Concurrent non-malignant co-morbidities that are uncontrolled
* History or symptoms indicative of brain or CNS metastases
* Prior diagnosis of any malignancy not cured by surgery alone less than 5 years before study entry (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Documented acute or chronic infection requiring antibiotic treatment
* Any concurrent chemo-, hormonal, immuno- or corticoid therapy
* Any prior chemotherapy for advanced or metastatic disease
* Any concurrent investigational treatment for advanced or metastatic disease
* History of relevant cardiovascular disease as follows:

  * Left ventricular ejection fraction (LVEF) below the institution's lower limit of normal, based on echocardiography (ECG) at rest
  * Uncontrolled or symptomatic congestive heart failure (New York Heart Association (NYHA) > 2
  * Uncontrolled or symptomatic arrhythmia and/or angina pectoris
  * Myocardial infarction during the last 2 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-03; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy measured by objective response rate (best response during the course of the study)

SECONDARY OUTCOMES:
Efficacy:
Clinical benefit rate
Duration of response
Time to progression (TTP)
Safety:
Incidence of adverse events (AEs)
Presence of human anti-murine antibodies after ertumaxomab infusion
Vital signs
Laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: José Baselga / Javier Cortes, Principal Investigator — Hospital Vall d'Hebron, Barcelona, Spain
Locations (5):
- Study Site, Austria
- Study Site, France
- Study Sites, Germany
- Study Site, Italy
- Barcelona, Spain

REFERENCES:
- [Background] Kiewe P, Hasmuller S, Kahlert S, Heinrigs M, Rack B, Marme A, Korfel A, Jager M, Lindhofer H, Sommer H, Thiel E, Untch M. Phase I trial of the trifunctional anti-HER2 x anti-CD3 antibody ertumaxomab in metastatic breast cancer. Clin Cancer Res. 2006 May 15;12(10):3085-91. doi: 10.1158/1078-0432.CCR-05-2436. PMID 16707606
- [Background] Zeidler R, Mysliwietz J, Csanady M, Walz A, Ziegler I, Schmitt B, Wollenberg B, Lindhofer H. The Fc-region of a new class of intact bispecific antibody mediates activation of accessory cells and NK cells and induces direct phagocytosis of tumour cells. Br J Cancer. 2000 Jul;83(2):261-6. doi: 10.1054/bjoc.2000.1237. PMID 10901380
- [Background] Zeidler R, Reisbach G, Wollenberg B, Lang S, Chaubal S, Schmitt B, Lindhofer H. Simultaneous activation of T cells and accessory cells by a new class of intact bispecific antibody results in efficient tumor cell killing. J Immunol. 1999 Aug 1;163(3):1246-52. PMID 10415020
- [Background] Ruf P, Lindhofer H. Induction of a long-lasting antitumor immunity by a trifunctional bispecific antibody. Blood. 2001 Oct 15;98(8):2526-34. doi: 10.1182/blood.v98.8.2526. PMID 11588051